CLINICAL TRIAL: NCT00586105
Title: A Multicenter Uncontrolled Study of Sorafenib in Patients With Unresectable and/or Metastatic Renal Cell Carcinoma
Brief Title: Phase III Study of Sorafenib in Patients With Renal Cell Carcinoma (RCC)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11559
Record Dates: First submitted 2007-12-21; First posted 2008-01-04 (Estimated); Results first posted 2010-10-01 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2014-03

CONDITIONS: Carcinoma, Renal Cell
Keywords: Sorafenib; Nexavar; Metastatic RCC; Renal Cell Carcinoma; Unresectable RCC
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sorafenib (Nexavar, BAY43-9006) (Experimental): 400 mg (2 tablets of 200 mg) of sorafenib per oral (PO) twice daily (BID)
  Interventions: Drug: Sorafenib (Nexavar, BAY43-9006)

INTERVENTIONS:
Drug: Sorafenib (Nexavar, BAY43-9006) — 400 mg (2 tablets of 200 mg) of sorafenib per oral (PO) twice daily (BID)

SUMMARY:
A multicenter uncontrolled study of sorafenib in patients with unresectable and/or metastatic renal cell carcinoma (RCC) to assess the pharmacokinetic profile, safety and tolerability, and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have a life expectancy of at least 12 weeks
* Patients, who suffer from unresectable and/or metastatic, measurable RCC histologically or cytologically documented. Patients with rare subtypes of RCC such as pure papillary cell tumor, mixed tumor containing predominantly sarcomatoid cells, Bellini carcinoma, medullary carcinoma, or chromophobe oncocytic tumors are excluded from study participation.
* Patients who have received not more than one prior systemic therapy for advanced disease which was completed at least 30 days prior to the first dose of study medication.
* Patients who have at least one uni-dimensional measurable lesion by Computed Tomography (CT)-scan or Magnetic Resonance Imaging (MRI) according to Response Evaluation Criteria in Solid Tumours (RECIST)
* Patients with "Intermediate" or "low" risk per the Motzer score
* Patients who have an Eastern Co-operative Oncology Group (ECOG) performance status of 0 or 1
* Adequate bone marrow, liver and renal function at screening as assessed by the following:
* Total bilirubin < 1.5 x the upper limit of normal.
* Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST) < 2.5 x upper limit of normal (< 5 x upper limit of normal for patients with liver involvement of their cancer).
* Amylase and lipase < 1.5 x the upper limit of normal.

  * Serum creatinine < 2.0 x the upper limit of normal.
  * Prothrombin Time (PT) or International Normalized Ratio (INR) and Partial Thromboplastin Time (PTT) < 1.5 x upper limit of normal

Exclusion Criteria:

* Previous or concurrent cancer that is distinct in primary sit or histology from the cancer being evaluated in this study EXCEPT cervical carcinoma in situ, adequately treated basal cell carcinoma, superficial bladder tumors [Ta (Noninvasive papillary carcinoma), Tis (Carcinoma in situ: "flat tumor") and T1 (Tumor invades subepithelial connective tissue)] or any cancer curatively treated > 3 years prior to study entry)
* Patients who completed their prior systemic treatment regimen less than 30 days
* Cardiac arrhythmias requiring anti-arrhythmic (excluding beta blockers or digoxin), symptomatic coronary artery disease or ischemia
* Active clinically serious bacterial or fungal infections
* Known history of human immunodeficiency virus (HIV) infection or chronic hepatitis B or C requiring current interferon treatment
* Symptomatic metastatic brain or meningeal tumors unless the patient is > 6 months from definitive therapy, has a negative imaging studies within 4 weeks of study entry and is clinically stable with respect to the tumor at the time of study entry.
* Patients with evidence or history of bleeding diathesis.
* Patients with seizure disorder requiring medication
* History of organ allograft
* Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
* Pregnant or breast-feeding patients.

Excluded concomitant medications:

* Concurrent anti-cancer chemotherapy, immunotherapy, or hormonal therapy except Bisphosphonates
* Radiotherapy during study or within 3 weeks of start of study drug.
* Biological response modifiers, such as Granulocyte-Colony Stimulating Factor (G-CFS) or Granulocyte macrophage colony-stimulating factor (GM-CFS), within 3 weeks prior to study entry or during study
* Significant surgery within 4 weeks prior to start of study drug
* Autologous bone marrow transplant or stem cell rescue within 4 months of study
* Investigational drug therapy during or within 4 weeks prior to first drug administration and during the study
* St John's Wort
* Xiao Chai Hu Tang
* Prior and concomitant use of Bevacizumab, and all other drugs (investigational or licensed) that target Vascular Endothelial Growth Factor (VEGF)/VEGF-Receptors, Raf-kinase inhibitors (RKI), Methyl Ethyl Ketone (MEK) or Farnesyl transferase inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2005-12; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (6):
- China (3):
  - Nanjing, Jiangsu
  - Beijing
  - Shanghai
- Taiwan (3):
  - Tainan, Tainan
  - Taipei
  - Taoyuan District

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were outpatients with histologically or cytologically confirmed, unresectable and/or metastatic, measurable clear Renal Cell Carcinoma (RCC) who had received not more than one prior systemic therapy. They were enrolled between 29 Dec 2005 and 29 Sep 2006 at 4 centers in China and 4 in Taiwan.
Pre-assignment Details: A total of 51 Asian subjects were enrolled in the trial. Twelve failed screening (11 protocol violations, 1 adverse event); the remaining 39 received at least 1 dose of study drug.
Period: Overall Study
Arm/Group | Sorafenib (Nexavar, BAY43-9006)
Started | 39
Completed | 0
Not Completed | 39
Not completed — Adverse Event | 4
Not completed — Death | 2
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 3
Not completed — Disease progression | 19
Not completed — Switched to commercial drug | 9
Not completed — Reason not reported | 1

BASELINE CHARACTERISTICS:
Arm/Group | Sorafenib (Nexavar, BAY43-9006)
Number analyzed (Participants) | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 30
Region of Enrollment [Number; unit: participants]
  Taiwan | 19
  China | 20
Eastern Cooperative Oncology Group (ECOG) Scale [Number; unit: participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status is a scale that measures how cancer affects a patient. The scale ranges from 0 (fully active) to 5 (dead). Subjects entering this study must have had an ECOG score of 0 or 1 (restricted in physically strenuous activity but ambulatory).
  participants
    ECOG 0 | 20
    ECOG 1 | 19
Motzer risk factors [Number; unit: participants] — The 5 Motzer risk factors correlate with overall survival in metastatic RCC. Patients with no factors (low-risk) have a favorable survival risk, patients with 1 or 2 risk factors survive a shorter time and constitute an intermediate-risk group, and those with 3 or more risk factors have the poorest survival and represent a poor-risk group.
  participants
    Low-risk (no risk factors) | 21
    Intermediate-risk (1 or 2 risk factors) | 18
Renal Cell Carcinoma subtype [Number; unit: participants] — Patients were categorized into 1 or 2 subgroups depending on the tumor histology: Clear cell or predominantly clear cell.
  participants
    Clear cell | 34
    Predominantly clear cell | 5
Time since first progression [Mean (Standard Deviation); unit: years] — Time since first progression was defined as the time from the first progression of the patient's disease after initial diagnosis until randomization into this study.
  years | 0.4 (0.6)
Time since initial diagnosis [Mean (Standard Deviation); unit: years] — Time since initial diagnosis was the mean time from initial diagnosis to randomization into the study.
  years | 1.7 (2.5)

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics Measured as Area Under Curve (AUC[0-12h])
Description: The AUC(0-12h) was the observed AUC, calculated using a combination of linear and log trapezoidal rules, from pre-dose to 12 hours post-dose. The normalized AUC (AUC norm) is AUC (0-12h) divided by (dose [mg]/weight [kg]).
Time Frame: 12 hours after at least 21 days of uninterrupted dosing
Population: A full pharmacokinetics (PK) profile was obtained in 32 of the 39 patients after at least 21 days of uninterrupted twice daily (BID) dosing.
Measure: Mean (Standard Deviation); unit: mg*hour/Liter
Arm/Group | Sorafenib (Nexavar, BAY43-9006)
Number analyzed (Participants) | 32
mg*hour/Liter
  AUC (0-12h) | 35.5 (16.1)
  AUC norm | 5.7 (3.0)

2. Primary Outcome: Pharmacokinetics Measured as Concentration (Cmax at Tmax and Cmin at Tmin)
Description: Cmax (maximum concentration) was measured at the time point at which the maximum concentration (Tmax) was observed. Cmin (minimum concentration) was measured at the time point at which the minimum concentration (Tmin) was observed.
Time Frame: 12 hours after at least 21 days of uninterrupted dosing
Population: A full PK profile was obtained in 32 of the 39 patients after at least 21 days of uninterrupted BID dosing.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Sorafenib (Nexavar, BAY43-9006)
Number analyzed (Participants) | 32
mg/L
  Cmax | 4.5 (2.4)
  Cmin | 2.0 (0.9)

3. Primary Outcome: Pharmacokinetics Measured as Concentration (Cmax Normalized at Tmax and Cmin Normalized at Tmin)
Description: Cmax (maximum concentration) was measured at the time point at which the maximum concentration (Tmax) was observed. Cmin (minimum concentration) was measured at the time point at which the minimum concentration (Tmin) was observed. The normalized variables (Cmax norm and Cmin norm) are the variables (Cmax and Cmin, see Primary Outcome Measure 2) divided by [dose (mg)/weight (kg)].
Time Frame: 12 hours after at least 21 days of uninterrupted dosing
Population: A full PK profile was obtained in 32 of the 39 patients after at least 21 days of uninterrupted BID dosing.
Measure: Mean (Standard Deviation); unit: Kg/L
Arm/Group | Sorafenib (Nexavar, BAY43-9006)
Number analyzed (Participants) | 32
Kg/L
  Cmax norm | 0.7 (0.5)
  Cmin norm | 0.3 (0.2)

4. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression-free survival (PFS) was defined as the time from the date of receipt of first dose of study drug to disease progression, radiological or clinical, or death, whichever was earlier. Subjects still alive without tumor progression at the time of analysis were censored at their date of last tumor evaluation.
Time Frame: Number of days from date of first dose of study drug to date first observed disease progression or death (whichever was earlier) was documented up to 17.25 months
Population: All subjects who received at least 1 dose of drug (the intent to treat [ITT] population) were included in the analysis. Thirty-nine patients received at least 1 dose of drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sorafenib (Nexavar, BAY43-9006)
Number analyzed (Participants) | 39
months | 5.5 [4.1 to 7.8]

5. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) was measured from the date of first dose of study drug until the date of death due to any cause. Survival time for subjects still alive at the time of analysis was censored at the date of last contact.
Time Frame: Time from start of therapy to death up to 17.25 months
Population: as for outcome 4
Measure: Median (Full Range); unit: months
Arm/Group | Sorafenib (Nexavar, BAY43-9006)
Number analyzed (Participants) | 39
months | 7.8 [0.9 to 13.4]

6. Secondary Outcome: Time to Progression (TTP)
Description: Time to progression (TTP) was defined as the time from date of receipt of first dose of study drug to disease progression, radiological or clinical. Subjects without tumor progression at the time of analysis were censored at their last date of tumor evaluation.
Time Frame: Time from start of study medication to clinical or radiological disease progression which ever occurs first up to 17.25 months
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sorafenib (Nexavar, BAY43-9006)
Number analyzed (Participants) | 39
months | 5.5 [4.1 to 7.4]

7. Secondary Outcome: Disease Control (DC)
Description: The DC was defined as subjects who had a best response rating of complete response (CR), partial response (PR), or stable disease (SD) according to Response Evaluation Criteria in Solid Tumors (RECIST) that was maintained for at least 28 days from the first demonstration of that rating. CR: disappearance of all clinical and radiological evidence of tumor (both target and non-target). PR: at least a 30% decrease in the sum of longest diameters (LD) of target lesions taking as reference the baseline sum LD. SD: steady state of disease; do not qualify for PR or progressive disease (PD).
Time Frame: From start to end of study medication up to 17.25 months
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Sorafenib (Nexavar, BAY43-9006)
Number analyzed (Participants) | 39
participants
  disease control | 32
  no disease control | 6
  not evaluated | 1

8. Secondary Outcome: Overall Best Response
Description: The best overall response was defined as the number of subjects with a confirmed CR, PR, SD, or PD. Tumor response was evaluated using RECIST. PD: at least a 20% increase in the sum of LD of measured lesions taking as ref. the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. Appearance of new lesions will also constitute PD. In exceptional circumstances, unequivocal progression of a non-measured lesion may be accepted as evidence of disease progression.
Time Frame: Best response observed from start to end of study medication up to 17.25 months
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Sorafenib (Nexavar, BAY43-9006)
Number analyzed (Participants) | 39
participants
  Complete Response (CR) | 0
  Partial Response (PR) | 5
  Stable Disease (SD) | 27
  Progressive Disease (PD) | 6
  not evaluated | 1

9. Secondary Outcome: Overall Response Duration
Description: Overall response duration was to be calculated for subjects who had a confirmed PR or CR, defined as the time from first assessment showing a PR or CR to progression or death.
Time Frame: From PR or CR to progression or death up to 17.25 months
Population: All subjects who received at least 1 dose of drug (the intent to treat [ITT] population) were included in the analysis. Thirty-nine patients received at least 1 dose of drug. The overall response duration was determined on the 5 subjects who had a PR.
Measure: Median (Full Range); unit: months
Arm/Group | Sorafenib (Nexavar, BAY43-9006)
Number analyzed (Participants) | 5
months | 7.4 [5.4 to 12.9]

10. Secondary Outcome: Time to Objective Response
Description: Time to objective response was defined as the time from the date of receipt of first dose of study drug to first assessment showing a confirmed PR or CR.
Time Frame: Time from start of study medication to first documented PR or CR up to 17.25 months
Population: All subjects who received at least 1 dose of drug (the intent to treat [ITT] population) were included in the analysis. Thirty-nine patients received at least 1 dose of drug. Time to objective response was determined on the 5 subjects who had a PR.
Measure: Median (Full Range); unit: months
Arm/Group | Sorafenib (Nexavar, BAY43-9006)
Number analyzed (Participants) | 5
months | 1.4 [1.3 to 18.3]

ADVERSE EVENTS:
Time Frame: From First Patient First Visit (FPFV) to Last Patient Last Visit (LPLV).
Description: Acronyms used: Gastrointestinal (GI), Genitourinary (GU), Not Otherwise Specified (NOS), Absolute Neutrophil Count (ANC), Aspartate aminotransferase (AST), Partial Thromboplastin Time (PTT), Alanine aminotransferase (ALT), Common Terminology Criteria for Adverse Events (CTCAE)
Arm/Group | Sorafenib (Nexavar, BAY43-9006)
Serious Adverse Events (participants affected / at risk) | 12/39
Other Adverse Events (participants affected / at risk) | 39/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib (Nexavar, BAY43-9006) (N=39)
Hemoglobin (Blood and lymphatic system disorders) | 1
Platelets (Blood and lymphatic system disorders) | 1
Anorexia (Gastrointestinal disorders) | 1
Obstruction, GI, Small Bowel NOS (Gastrointestinal disorders) | 1
Fever (General disorders) | 3
Pain, Abdomen NOS (General disorders) | 1
No Code In CTCAE (General disorders) | 3
Infection With Normal ANC, Biliary Tree (Infections and infestations) | 1
Infection With Normal ANC, Paranasal (Infections and infestations) | 1
Infection With Normal ANC, Urinary Tract NOS (Infections and infestations) | 1
Infection With Unknown ANC, Skin (Cellulitis) (Infections and infestations) | 1
Fracture (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary - Other (Respiratory, thoracic and mediastinal disorders) | 2
Hand-Foot Skin Reaction (Skin and subcutaneous tissue disorders) | 1
Hemorrhage, GI, Duodenum (Vascular disorders) | 1
Hemorrhage - Other (Vascular disorders) | 1
Hemorrhage Pulmonary, Bronchus (Vascular disorders) | 1
Hemorrhage, GU, Urinary NOS (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib (Nexavar, BAY43-9006) (N=39)
Hemoglobin (Blood and lymphatic system disorders) | 9
PTT (Blood and lymphatic system disorders) | 3
Edema: Limb (Blood and lymphatic system disorders) | 4
Supraventricular Arrhythmia, Sinus Tachycardia (Cardiac disorders) | 2
Hypertension (Cardiac disorders) | 7
Tinnitus (Ear and labyrinth disorders) | 4
Anorexia (Gastrointestinal disorders) | 11
Constipation (Gastrointestinal disorders) | 9
Diarrhea (Gastrointestinal disorders) | 14
Distension (Gastrointestinal disorders) | 3
Mucositis (Functional/Symptomatic), Oral Cavity (Gastrointestinal disorders) | 3
Mucositis (Clinical Exam), Oral Cavity (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 3
GI - Other (Gastrointestinal disorders) | 2
Periodontal (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 5
Fever (General disorders) | 5
Weight Gain (General disorders) | 2
Insomnia (General disorders) | 2
Fatigue (General disorders) | 12
Weight Loss (General disorders) | 9
Pain, Back (General disorders) | 5
Pain, Chest/Thorax NOS (General disorders) | 2
Pain, Chest Wall (General disorders) | 2
Pain, Dental/Teeth/Peridontal (General disorders) | 2
Pain, Extremity - Limb (General disorders) | 2
Pain, Abdomen NOS (General disorders) | 5
Pain, Head/Headache (General disorders) | 3
Pain, Joint (General disorders) | 5
Pain, Bone (General disorders) | 7
Pain, Other (General disorders) | 2
Pain, Stomach (General disorders) | 4
Flu-Like Syndrome (General disorders) | 3
Infection With Normal ANC, Urinary Tract NOS (Infections and infestations) | 2
Infection - Other (Infections and infestations) | 2
Infection With Unknown ANC, Skin (Cellulitis) (Infections and infestations) | 2
Alkaline Phosphatase (Metabolism and nutrition disorders) | 2
ALT (Metabolism and nutrition disorders) | 7
Amylase (Metabolism and nutrition disorders) | 2
AST (Metabolism and nutrition disorders) | 8
Creatinine (Metabolism and nutrition disorders) | 4
Bilirubin (Hyperbilirubinemia) (Metabolism and nutrition disorders) | 6
Hypercalcemia (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hyperuricemia (Metabolism and nutrition disorders) | 8
Hypoalbuminemia (Metabolism and nutrition disorders) | 5
Lipase (Metabolism and nutrition disorders) | 5
Hypophosphatemia (Metabolism and nutrition disorders) | 9
Metabolic/Lab - Other (Metabolism and nutrition disorders) | 6
Arthritis (Musculoskeletal and connective tissue disorders) | 2
Dizziness (Nervous system disorders) | 2
Incontinence, Urinary (Renal and urinary disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 11
Nasal/Paranasal Reactions (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (Shortness Of Breath) (Respiratory, thoracic and mediastinal disorders) | 3
Voice Changes (Respiratory, thoracic and mediastinal disorders) | 5
Acne (Skin and subcutaneous tissue disorders) | 6
Alopecia (Skin and subcutaneous tissue disorders) | 14
Hand-Foot Skin Reaction (Skin and subcutaneous tissue disorders) | 25
Pruritus (Skin and subcutaneous tissue disorders) | 6
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 9
Flushing (Skin and subcutaneous tissue disorders) | 3

LIMITATIONS AND CAVEATS:
The median for ´Overall Survival (OS)´ and the median for ´Overall Response Duration´ reported are the median of each distribution including the censored data. The correct estimates of these medians were not evaluable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less